CLINICAL TRIAL: NCT04249661
Title: Differential Effects of Bacteria Colonising Venous Leg Ulcers on Pain and Healing Rates
Status: Completed | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Professor Eamon Kavanagh Prinicipal Investigator, University Hospital of Limerick
Other Study IDs: DVS003
Record Dates: First submitted 2020-01-16; First posted 2020-01-31 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Wound swabs will be obtained from the venous leg ulcer from participants and sent to the Microbiology lab for culture and sensitivity testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Study aims to identify whether venous leg ulcers which are colonised by Pseudomonas Aeruginosa cause more pain than those which are not and if this bacteria affects healing time. This may determine how venous ulcer infections are treated in order to improve symtomatology and quality of life for patients with these chronic wounds.

DETAILED DESCRIPTION:
Pseudomonas is a gram-negative bacillus which commonly colonises lower limb venous ulcers. It produces exotoxins and elastase as well as forming biofilms within chronic wounds.

Its effects on venous ulcer healing are debated. The objective of this study is to examine the effects on Pseudomonas Aeruginosa colonisation on the pain expereinces and healing rates of venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. All patients age 18+ with lower limb venous ulcers as diagnosed on clinical history and examination.
2. Are willing and capable to voluntarily sign a statement of informed consent to take part in this study.
3. With an ABPI of >/= 0.8 and/or palpable pedal pulses on clinical exam.
4. Without evidence (either clinical or diagnostic) of other causes of lower limb ulceration, namely vasculitis, local dermopathology, congenital syndromes or arterial insufficiency (see above).
5. If equipoise or disagreement between two independent clinicians exist, The ultimate decision as to inclusion/exclusion will be made by the P.I

Exclusion Criteria:

1. Patients unable to provide informed consent.
2. Patients under the age of 18
3. Patients with arterial insufficiency manifesting as ABPI's of <0.8
4. Known or suspected alternate likely primary cause of lower limb ulceration (vasculitis, dermatological disease, underlying congenital syndrome).
5. Patients who are deemed unsuitable due to any circumstances as deemed appropriate by the P.I.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular patients with new and old venous ulcers to their lower limbs. As deemed suitable as per the inclusion/exclusion criteria. As deemed suitable by the P.I.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Pain burden of venous ulcers colonised by Pseudomonas Aeruginosa | 1 year
  Pain will be examined with respect to underlying microbiota detected by wound culture and sensitivity. The Brief Pain Inventory (Short Form) will be used for assessment purposes.
Presentations and Admissions | 1 year
  Rates of re-presentation for treatment with respect to underlying wound culture and sensitivity. Number of patient visits to the Vascular Clinic for treatment will be measured.

SECONDARY OUTCOMES:
Analgesia Requirements | 1 year
  Number of participants with pain requiring analgesia will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eamon Kavanagh, MD FRCSI, Principal Investigator — University Hospital of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided